CLINICAL TRIAL: NCT02697292
Title: A Randomized Double Blind Placebo Controlled Study of Intravenous Immunoglobulin (IVIG) Patients With Voltage Gated Potassium Channel Complex (VGKC) Antibody Associated Autoimmune Epilepsy
Brief Title: IVIG in Patients With VGKC Ab Associated Autoimmune Epilepsy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Grifols Shared Services North America (Unknown); Option Care (Industry)
Responsible Party: Principal Investigator, Sean Pittock, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-005649
Record Dates: First submitted 2016-02-19; First posted 2016-03-03 (Estimated); Results first posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Autoimmune Epilepsy
Keywords: Intravenous Immunoglobulin; VGKC; Autoimmune epilepsy; Gamumex-C
MeSH Terms: interventions — Immunoglobulins, Intravenous; Hizentra; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo/Normal Saline Group (Placebo Comparator): Subjects will receive placebo for 4 infusions. After completion of the blinded phase, subjects will receive IVIG for 4 infusions. Subjects will maintain their stable dose of antiepileptic meds.
  Interventions: Drug: Intravenous Immunoglobulin; Drug: Placebos; Drug: Normal Saline
- Intravenous Immunoglobulin (IVIG) (Gamunex-C) Group (Active Comparator): Subjects will receive IVIG for 4 infusions. Subjects will maintain their stable dose of antiepileptic meds.
  Interventions: Drug: Intravenous Immunoglobulin; Drug: Normal Saline

INTERVENTIONS:
Drug: Intravenous Immunoglobulin — GAMUNEX-C is a clear a ready-to-use sterile solution of human immune globulin protein for intravenous administration. Dose will be determined based on ideal wt. with not to exceed 80 grams. Subjects will receive 0.5g/kg daily for 1 day [week 1 day 1], then will receive 1g/kg not exceeding 80 grams daily for 1 day [week 1 day 2]. Then once every 2 weeks subjects will receive 0.6g/kg IVIG for 4 weeks [week 3 and 5] for 2 infusions.
  Other Names: Gamunex-C
Drug: Placebos — Normal Saline is a sterile, nonpyrogenic solution for fluid and electrolyte replenishment. Dose will be determined based on ideal wt. with not to exceed 80 grams. Dose will be determined based on ideal wt. with not to exceed 80 grams. Subjects will receive 0.5g/kg daily for 1 day [week 1 day 1], then will receive 1g/kg not exceeding 80 grams daily for 1 day [week 1 day 2]. Then once every 2 weeks subjects will receive 0.6g/kg for 4 weeks [week 3 and 5] for 2 infusions.
  Other Names: Normal Saline
  Arms: Placebo/Normal Saline Group
Drug: Normal Saline — Normal Saline is a sterile, nonpyrogenic solution for fluid and electrolyte replenishment. Subjects will receive 500 ml normal saline before and after the higher dose infusion of 1g/kg

SUMMARY:
The purpose of this study is to determine whether intravenous immunoglobulin (IVIG) treatment reduces significantly the number of epileptic seizures in cases of autoimmune epileptic seizures.

DETAILED DESCRIPTION:
The purpose of this study is to determine if intravenous immunoglobulin (IVIG) treatment significantly reduces the number of epileptic seizures in cases of autoimmune epilepsy. Potential participants will be screened at an outpatient neurology clinic visit appointment. Interested qualified potential participants will be consented and offered participation in this trial. Once consent has been obtained, and it is determined that the participant meets all inclusion criteria, the participant will be randomized to either IVIG or placebo treatment for the next 5 weeks. Participants will return to Mayo Clinic for an evaluation. Those participants that received the placebo for 5 weeks will be given IVIG in an open label fashion for 5 weeks (week 7-11) then return to Mayo Clinic for evaluation. All participants will receive monthly phone calls after they complete the IVIG treatment for a period of 1 year from the end of IVIG 5 week course.

ELIGIBILITY:
Inclusion Criteria:

* Seropositivity for Voltage Gated Potassium Channel Complex (VGKC) complex antibodies or positive for Leucine-Rich, Glioma Inactivated 1 (LGI1)/contactin-associated protein-like 2 (CASPR2) Antibody by cell based assay.
* And ≥ 2 seizures per week (mean of total over 1 week)
* And duration of epilepsy <3 years
* Male or female between the ages of 18 and 80 years of age
* Women and men of child bearing potential must agree to use a reliable form of contraception throughout the course of the study.
* Homecare treatment agency available at place of residence.

Exclusion Criteria:

* History of thrombotic episodes within the 2 years prior to enrollment
* Known allergic or other severe reactions to blood products including intolerability to previous IVIG
* Immunoglobulin A (IgA) deficiency
* Prior failed trial of high dose steroid (prednisone >60mg daily or methylprednisolone >1g weekly for >2 weeks)
* Reproductive status:

  * Women who are pregnant,
  * Women who are breastfeeding,
  * Women and men of childbearing potential who are unwilling or unable to use an acceptable method of birth control to avoid pregnancy for the entire study period, as evaluated by the investigator. (Women of non-childbearing potential are those that have a history of hysterectomy, bilateral oophorectomy, or are postmenopausal with no history of menstrual flow for > 12 months prior to screen visit.)
* Any surgical procedure (except for minor surgeries) within 4 weeks prior to baseline.
* Evidence of serious uncontrolled concomitant diseases that may preclude patient participation (physician determined), as described; Other nervous system disease, cardiovascular disease, hematologic/hematopoiesis disease, respiratory disease, muscular disease, endocrine disease, renal/urologic disease, digestive system disease, congenital or acquired severe immunodeficiency
* Known active infection (excluding fungal infections of nail beds or caries dentium) within 4 weeks prior to baseline.
* Evidence of chronic active hepatitis B or C.
* Active ischemic heart disease in the past year prior to baseline.
* Patients should not have severe renal or hepatic disease (determined by treating physician).
* Severe hypertension

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-02; Primary Completion 2018-12-03 (Actual); Study Completion 2018-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean Pittock, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials.
- See also: PubMed — https://www.ncbi.nlm.nih.gov/pubmed/?term=Randomized+Placebo+Controlled+Trial+of+IVIG+in+autoimmune+LGI1%2FCASPR2+epilepsy

RESULTS

PARTICIPANT FLOW:
Groups:
- Intravenous Immunoglobulin (IVIG) (Gamunex-C) Group: Subjects who received IVIG for 4 infusions. Subjects maintained their stable dose of antiepileptic meds.
Period: Overall Study
Arm/Group | Placebo/Normal Saline Group | Intravenous Immunoglobulin (IVIG) (Gamunex-C) Group
Started | 9 | 8
Completed | 9 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Normal Saline Group | Intravenous Immunoglobulin (IVIG) (Gamunex-C) Group | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 70 [59 to 77] | 70 [66 to 77] | 70 [59 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 6 | 6 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Change in Seizure Frequency From Baseline to 5 Weeks
Description: The number of subjects who experience a ≥ 50% reduction in seizure frequency
Time Frame: baseline, 5 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Normal Saline Group | Intravenous Immunoglobulin (IVIG) (Gamunex-C) Group
Number analyzed (Participants) | 9 | 8
Participants | 2 | 6
Statistical Analysis 1: Comparison: Placebo/Normal Saline Group vs Intravenous Immunoglobulin (IVIG) (Gamunex-C) Group; Test type: Superiority; p = 0.044, t-test, 1 sided; Odds Ratio (OR) = 10.5, 95% CI 2-sided [1.1 to 98.9]

2. Secondary Outcome: Change in Cognitive Assessment
Description: Number of subjects who experienced stable or improved cognitive assessment. Cognitive status was measured using the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS). The RBANS is a individually administered standardized battery of 12 tests that measure cognitive decline or improvement taking approximately 30 minutes. Five index scores are computed from the RBANS (immediate memory, language, visuospatial, attention, delayed memory) that are combined to provide the Total Score (range 40-160)
Time Frame: baseline, 5 weeks
Population: One subject did not complete the assessment at week 5 for the placebo arm
Measure: Count of Participants; unit: Participants
Groups:
- Intravenous Immunoglobulin (IVIG) (Gamunex-C) Group: Subjects who received IVIG for 4 infusions. Subjects will maintain their stable dose of antiepileptic meds.
Arm/Group | Placebo/Normal Saline Group | Intravenous Immunoglobulin (IVIG) (Gamunex-C) Group
Number analyzed (Participants) | 8 | 8
Participants | 5 | 8
Statistical Analysis 1: Comparison: Placebo/Normal Saline Group vs Intravenous Immunoglobulin (IVIG) (Gamunex-C) Group; Test type: Superiority; p = 0.100, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: The study period during which adverse events were collected is defined as the period from the initiation of any study procedures to the end of the study treatment follow-up, approximately 6 weeks.
Arm/Group | Placebo/Normal Saline Group | Intravenous Immunoglobulin (IVIG) (Gamunex-C) Group
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 4/9 | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/Normal Saline Group (N=9) | Intravenous Immunoglobulin (IVIG) (Gamunex-C) Group (N=8)
Encephalitis (Nervous system disorders) | 1 (1) | 0 (0)
Fall (General disorders) | 1 (1) | 1 (1)
Headache (General disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-09): https://cdn.clinicaltrials.gov/large-docs/92/NCT02697292/Prot_SAP_000.pdf